CLINICAL TRIAL: NCT02306499
Title: Outcome of ICSI Using Cryopreserved Testicular Sperm From Infertile Men With Varicocele-associated Azoospermia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Al-Hussini Jad Abdel-latif, M.B.B.Ch., Egypt - Sohag - Nasser City - Sohag University - Faculty Of Medicine - Dermatology, Venereology and Andrology Department, Sohag University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 729/2014; 729/259/2014 (Other: Sohag University - Faculty of Medicine)
Record Dates: First submitted 2014-11-22; First posted 2014-12-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-11

CONDITIONS: ICSI AZOOSPERMIA VARICOCELE
Keywords: VARICOCELE-AZOOSPERMIA-ICSI
MeSH Terms: interventions — Sperm Injections, Intracytoplasmic

ARMS (2):
- ICSI WITH CRYOPRESERVED SPERM FROM NOA WITH VARICOCELE (Experimental): ICSI cases using cryopreserved testicular sperm from infertile azoospermic men, with proven diagnosis of varicocele (clinical & sonographic), which will be used for ICSI in an ART program
  Interventions: Procedure: ICSI
- ICSI WITH CRYOPRESERVED SPERM FROM NOA WITH NO VARICOCELE (Experimental): ICSI cases using cryopreserved testicular sperms from infertile azoospermic men due to etiologies other than varicocele
  Interventions: Procedure: ICSI

INTERVENTIONS:
Procedure: ICSI — Intracytoplasmic Sperm Injection

SUMMARY:
This study will include cryopreserved sperm from infertile azoospermic men, with proven diagnosis of varicocele (clinical & sonographic), which will be used for ICSI in an ART program in Sohag. Patients personal and medical history and socio-demographic data will be retrieved from their saved medical files.

DETAILED DESCRIPTION:
Study approval: The study will be submitted for approval by Research and Ethical committees at Faculty of Medicine, Sohag University.

This study will include cryopreserved sperm from infertile azoospermic men, with proven diagnosis of varicocele (clinical & sonographic), which will be used for ICSI in an ART program in Sohag .

Patients personal and medical history and socio-demographic data will be retrieved from their saved medical files.

Study design: Prospective, controlled clinical study. Control group: ICSI cases using cryopreserved sperms from infertile azoospermic men due to etiologies other than varicocele. Cases with known female factor infertility will be excluded.

Outcome Measures: fertilization rate, embryo quality, chemical pregnancy and clinical pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* cryopreserved sperm from infertile azoospermic men, with proven diagnosis of varicocele (clinical & sonographic), which will be used for ICSI in aى ART program.
* ICSI cases using cryopreserved sperms from infertile azoospermic men due to etiologies other than varicocele.

Exclusion Criteria:

* Cases with known female factor infertility

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-05 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy: documentation of gestational sac and fetal pulsation by transvaginal US 15 days after B-HCG assessment. | 6/2014 up to one year.

SECONDARY OUTCOMES:
Fertilization Rate: percentage of fertilized oocyte. | 6/2014 up to one year.
Embryo Quality: morphological assessment of the developing embryo. | 6/2014 up to one year.
Chemical pregnancy: B-human chorionic gonadotropin (B-HCG) at day 15 after embryo transfer. | 6/2014 up to one year.

CONTACTS AND LOCATIONS:
Overall Officials: Ramadan Saleh, MD, Study Director — Sohag University; Reham Ezz-Eldawla, MD, Study Director — Sohag University; Mohamed Yahya, MD, Study Director — Sohag University; Muhammed Fawzy, Study Director — Ibn Sina Hospital
Locations (1):
- Ajyal Hospital, Sohag, Egypt